CLINICAL TRIAL: NCT00460889
Title: Renal Donor Comparison of Outcomes: Hand Assist Versus Laparoscopic Nephrectomy
Status: Withdrawn | Type: Observational
Why Stopped: Principal Investigator left institution
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAB9478
Record Dates: First submitted 2007-04-13; First posted 2007-04-17 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Living Renal Donor
Keywords: hand assist; laparoscopy; renal donor; outcomes

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: donor nephrectomy — The objective of this protocol is to look at the outcomes of laparoscopic donor nephrectomy performed by using hand assisted (HA)or entirely laparoscopic (LDN) surgical techniques. To define the advantages of each technique, we will use records of patients who underwent laparoscopic live kidney donation with HALDN.

SUMMARY:
This study is designed to look at outcomes of patients who have undergone hand assisted laparoscopic donor nephrectomy versus totally laparoscopic donor nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* any person undergoing minimally invasive donor nephrectomy surgery at NewYork Hospital/Columbia.

Exclusion Criteria:

* any person undergoing open donor nephrectomy surgery at NewYork Hospital/Columbia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgical clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Prevalence of postoperative comfort and hospital stay satisfaction with HALDN | 1 week
Prevalence of postoperative comfort and hospital stay satisfaction with LDN | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Dennis L Fowler, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University College of Physicians and Surgeons, New York, New York, United States